CLINICAL TRIAL: NCT06643338
Title: Development of a Deep Learning System for Identification of Neuro-Ophthalmological Conditions on Color Fundus Photographs in Emergency Department
Acronym: DEEP-VISION
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: DMA_2024_6
Record Dates: First submitted 2024-08-09; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In recent years, artificial intelligence (AI) has been widely integrated into the medical field, contributing in particular to improved patient diagnosis. The BONSAI study, Brain and Optic Nerve Study with AI, in which our team is participating, has successfully demonstrated the ability of AI to identify individual neuro-ophthalmological or neurological pathologies affecting the optic nerves and/or brain, from a simple fundus image.

While this is a promising advance, it remains limited in current clinical practice. Our major challenge is to be able to identify a wider range of optic nerve and/or brain pathologies simultaneously in the same analysis, so as to improve patient management, especially for those referred to emergency departments. Indeed, in the absence of a precise diagnosis, complications can be irreversible and life-threatening.

Among the most alarming clinical signs in the emergency department is papilledema of stasis, which, accompanied by acute headaches, may indicate the presence of intracranial hypertension, inflammatory or ischemic pathology. The latter may be a manifestation of Horton's disease. Our team has developed an AI algorithm to diagnose retinal and optic nerve abnormalities based on retinophotographs taken under ideal conditions during scheduled consultations, and not on images of patients presenting to the emergency department. In hospitals without ophthalmology emergency departments, it is essential that emergency physicians (emergency physicians, general practitioners, neurologists) are able to assess the fundus in the absence of an ophthalmology specialist. This assessment, although part of the general examination, often presents challenges for non-ophthalmologists. The aim of our study is to improve the performance of our AI algorithm so that it can discriminate between different retinal and optic nerve pathologies in the emergency department. We therefore plan to build a database of fundus images by prospectively including patients presenting to the ophthalmology and neurology emergency departments of the Fondation Adolphe de Rothschild Hospital. The performance of the algorithm developed will be evaluated according to standard criteria of sensitivity, specificity, area under the curve (AUC) and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Presenting to the emergency department of the Fondation Adolphe de Rothschild hospital
* Express consent to participate in the study
* Member or beneficiary of a social security scheme

Exclusion Criteria:

* Patient under legal protection
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the emergency department of the Fondation Adolphe de Rothschild hospital with no signs of infection and/or ocular allergy (runny eye, red eye).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of correct predictions among all positive predictions out of all total predictions of the algorithm (positive + negative) | Day 30
  The gold standard will be the diagnosis made by a senior ophthalmologist on the basis of the patient's medical records consulted at D30 after the emergency visit

SECONDARY OUTCOMES:
Sensitivity of the algorithm for each eye disease | Day 30
  The gold standard will be the diagnosis made by a senior ophthalmologist on the basis of the patient's medical records consulted at D30 after the emergency visit
Specificity of the algorithm for each eye disease | Day 30
  The gold standard will be the diagnosis made by a senior ophthalmologist on the basis of the patient's medical records consulted at D30 after the emergency visit
Area under the curve (AUC) for each eye disease | Day 30
  The gold standard will be the diagnosis made by a senior ophthalmologist on the basis of the patient's medical records consulted at D30 after the emergency visit

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No